CLINICAL TRIAL: NCT01699256
Title: Enhanced Implementation of Low Back Pain Guidelines in General Practice: A Cluster Randomized Trial
Brief Title: Enhanced Implementation of Low Back Pain Guidelines in General Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008-58-0028
Record Dates: First submitted 2012-09-13; First posted 2012-10-03 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2015-07

CONDITIONS: Low Back Pain
Keywords: General Practice; Low Back Pain; Guideline; Health Plan Implementation; Referral and Consultation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced strategy (Experimental): Enhanced implementation strategy
  Interventions: Behavioral: Enhanced guideline implementation strategy
- Strategy as usual (Active Comparator): Normal implementation strategy
  Interventions: Behavioral: Guideline implementation as usual

INTERVENTIONS:
Behavioral: Guideline implementation as usual — Newsletters and Invitation to Meetings
  Arms: Strategy as usual
Behavioral: Enhanced guideline implementation strategy — Enhanced guideline implementation strategy
  Arms: Enhanced strategy

SUMMARY:
The aim of this study is to evaluate whether an enhanced strategy of implementation of the new guideline will lower the number of patients getting referred to secondary care spine centres compared to a normal implementation strategy.

DETAILED DESCRIPTION:
Introduction:

There is a need for more knowledge on how to introduce new guidelines effectively in general practice. A new low back pain treatment guideline is implemented in Denmark. This guideline demands that patients with low back pain who have not improved after eight weeks of primary care treatment should be referred to a secondary care spine centre.

Methods:

This is a cluster randomized trial. One hundred general practices define clusters and are randomly allocated to enhanced or usual implementation of the new guideline. The practices are all situated in the North Denmark Region and count two hundred general practitioners (GPs).

General practices in the control group will receive normal implementation of the new guideline, which include newsletters and briefings. In contrast the intervention group will receive an enhanced implementation strategy, adding visits from a consultant, two different stratification tools and feedback on guideline compliance. The two stratification tools: The STarT back screening tool (STarT) and a "Social and Occupational Screening" tool (SOS). The two screening tools subgroups patients and aids the clinicians in their choice of treatment.

Discussion:

To evaluate how change in behaviour may improve guideline adherence and patient treatment we plan two Ph.d. studies in relation to this study; one focusing on the clinical and an one on the economic aspects of the study. In addition a qualitative study is planned for patients refered to specialists in social medicine.

ELIGIBILITY:
Inclusion Criteria:

* Provider number in the North Denmark Region (Practice level)
* ICPC coded: L02, L03, L84, and L86 (Patient level)
* Age 18-65 years (Patient level)

Exclusion Criteria:

* No signed written consent form (Practice level)
* Earlier participation in project testing (Practice level)
* Already included (Patient level)
* Patients with "red flags"/signs of serious pathology (Patient level)
* Pregnancy (Patient level)
* Insufficient Danish language skills (Patient level)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1101 (Actual)
Dates: Start 2012-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Referral of patients to a secondary care back centre | 12 weeks

SECONDARY OUTCOMES:
Cost-effectiveness | 4, 8, and 52 weeks
Roland Morris 23q disability score | 4, 8, and 52 weeks
Numerical pain rating | 4, 8, and 52 weeks
EQ-5D (Life quality) | 4, 8, and 52 weeks
Sick-leave | 4, 8, and 52 weeks
Employment status | 4, 8, and 52 weeks

OTHER OUTCOMES:
Guideline compliance | During study
Actual delivered intervention | During study
Association between the STart Bact Tool and the functional disability | 8 weeks
  An ancillary analysis of the predictive ability of the STarT Back Tool

CONTACTS AND LOCATIONS:
Overall Officials: Allan Riis, Master, Principal Investigator — University of Aarhus
Locations (1):
- Research Unit for General Practice in the North Denmark Region, Aalborg, Aalborg, Denmark

REFERENCES:
- [Derived] Riis A, Rathleff MS, Jensen CE, Jensen MB. Predictive ability of the start back tool: an ancillary analysis of a low back pain trial from Danish general practice. BMC Musculoskelet Disord. 2017 Aug 23;18(1):360. doi: 10.1186/s12891-017-1727-6. PMID 28835238
- [Derived] Riis A, Jensen CE, Bro F, Maindal HT, Petersen KD, Bendtsen MD, Jensen MB. A multifaceted implementation strategy versus passive implementation of low back pain guidelines in general practice: a cluster randomised controlled trial. Implement Sci. 2016 Oct 21;11(1):143. doi: 10.1186/s13012-016-0509-0. PMID 27769263
- [Derived] Jensen CE, Riis A, Pedersen KM, Jensen MB, Petersen KD. Study protocol of an economic evaluation of an extended implementation strategy for the treatment of low back pain in general practice: a cluster randomised controlled trial. Implement Sci. 2014 Oct 8;9:140. doi: 10.1186/s13012-014-0140-x. PMID 25293975
- [Derived] Riis A, Jensen CE, Bro F, Maindal HT, Petersen KD, Jensen MB. Enhanced implementation of low back pain guidelines in general practice: study protocol of a cluster randomised controlled trial. Implement Sci. 2013 Oct 20;8:124. doi: 10.1186/1748-5908-8-124. PMID 24139140